CLINICAL TRIAL: NCT03854214
Title: Cortical Functional Connectivity as an Early Biomarker of Recovery in Spinal Cord Injury (Study 239481)
Brief Title: Investigation of Brain Functional MRI as an Early Biomarker of Recovery in Individuals With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Ann Choe, Assistant Professor, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 00182576; R21NS104644 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-02-26 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; MRI, Functional; Rehabilitation; Neuronal Plasticity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The study will be performed as a randomized, parallel group trial to determine if the amount of changes in brain functional connectivity outcome measures (i.e., between network connectivity) is significantly different between the group of patients that perform FES cycling and another group of patients that perform passive (sham) cycling.
  Official screening will be performed after participants consent by signing the study's consent form. Participants will be randomized into 2 groups: FES cycling (Group 1; n=24) and passive cycling (Group 2; n=24). The participants will undergo either an FES cycling or a passive cycling sessions for 4 weeks, 3 times a week. MRI will be performed on all participants at the beginning (prior to cycling sessions) and at the end of the 2nd and 4th weeks of the intervention program. ISNCSCI evaluations will be performed to coincide with the dates of MRI acquisitions, to determine the neurological level and the degree of sensory and motor impairments.
Who Masked: Participant, Care Provider
Masking Description: This study is a double-blinded randomized trial. Study physicians and research staff who perform study measurements on participants will be blinded from the intervention the study participants receive. Study participants will not be informed of the intervention he/she will receive. However, because of the nature of the interventions, study participant cannot be completely blinded to the treatment they will receive, as some participants may have residual motor and sensory functions and 'feel' which intervention they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Functional Electric Stimulation cycling (Active Comparator): The Functional Electrical Stimulation (FES) cycling group will use RT300 ergometer (Restorative Therapies, Inc) with stimulation on.
  Interventions: Device: Functional Electric Stimulation cycling
- Passive Cycling (Sham Comparator): The passive cycling group will use the same RT300 ergometer with stimulation off.
  Interventions: Device: Passive cycling

INTERVENTIONS:
Device: Functional Electric Stimulation cycling — The Functional Electrical Stimulation (FES) cycling group will use RT300 ergometer (Restorative Therapies, Inc). Bilateral glutei, quadriceps and hamstrings will be stimulated. The stimulation parameters will be set as follows: waveform biphasic, charged balanced; phase duration of 250 microseconds; pulse rate 33-45 pps. The stimulus intensity will be adjusted for individual patients and muscle group so that a tolerable stimulation is provided that will generate a cycling action. Target cycling speed is 50 revolutions per minute (RPM). Resistance will be automatically adjusted by the FES bike according to the subject's performance. When fatigue occurs, participants will continue cycling with electrical stimulation and motor support. FES therapy will be administered for one hour per session 3 times a week.
  Other Names: RT300 ergometer
  Arms: Functional Electric Stimulation cycling
Device: Passive cycling — The passive cycling group will use the same RT300 ergometer however during this period stimulation will not be turned on. Instead, continuous motor support will be activated resulting in passive cycling. Target cycling speed is 50 RPM. Participants assigned to passive cycling will be required to have one hour of passive therapy 3 times a week for the entire duration of treatment assignment.
  Other Names: RT300 ergometer
  Arms: Passive Cycling

SUMMARY:
Early detection of response to therapeutic intervention is vital, as it will enable early termination of intervention in non-responding patients, prevent unnecessary financial burden, and allow for early changes to the intervention program. Previous functional MRI (fMRI) studies have shown that changes in brain functional network in spinal cord injury (SCI) patients can occur after as little as one week of intervention. Resting state fMRI (rsfMRI) is a type of fMRI that does not require performance of explicit motor tasks, which makes the method especially suitable for SCI patient population. In this project, the investigators propose that rsfMRI outcome measures can be used to detect early brain functional network changes that occur during intervention, and that the changes will be predictive of recovery in chronic SCI patients.

DETAILED DESCRIPTION:
Early detection of response to spinal cord injury (SCI) therapeutic intervention programs is vital, as it will enable early termination of intervention in non-responding patients, prevent unnecessary financial burden, and allow for early changes of the programs. In this project, the investigators propose that resting state functional MRI (rsfMRI) can be used to detect early brain functional network changes that occur during intervention, and that the changes will be predictive of recovery in chronic SCI patients. The long-term goal of this study is to establish rsfMRI as a new imaging biomarker that is predictive of progress towards recovery in response to therapy. International Standard of Neurological Classification for Spinal Cord Injury (ISNCSCI) scoring system is the most widely used clinical classification system of SCI that describes neurological injury level and degree of functional preservation. It is also used to monitor the progress and response to interventions such as functional electrical stimulation (FES) therapy. However, monitoring responses using ISNCSCI is challenging, because its ability to describe the degree of functional loss is limited. Therefore, there is a need in the field of SCI for a biomarker that is more sensitive to changes in function. The investigators will recruit 2 groups of 24 chronic SCI patients. In one group, the investigators will characterize the baseline time profile of rsfMRI outcome measures acquired during a 4-weeks passive cycling program, where movement is driven only by the cycle's motor (no electric stimulation). RsfMRI data of the patients acquired at weeks 0, 2, and 4 will be used perform functional parcellation of the sensorimotor cortex using independent component analysis (ICA) and spectral clustering analysis (SCA) approaches. BNC will be calculated between pairs of sensory and motor brain parcels. Sensory and motor ISNCSCI scores will also be measured at weeks 0, 2, and 4. The investigators will then test the hypothesis that the investigators will observe stable baseline measures of sensory and motor cortex BNC and ISNCSCI scores of the patients during the 4-week passive cycling program, with minimal to no change in values. In the second group, the investigators will characterize the time profile of the cortical reorganization in chronic SCI patients that occurs during the four-week FES cycling. Specifically, the investigators predict that the investigators will observe early functional network changes in the sensorimotor cortex of SCI patients (measured using BNC) at week 2 of the four-week FES cycling program, which will be predictive of changes in ISNCSCI scores (neurological outcomes) at week 4. Finally, the longitudinal intra-subject reproducibility of the two parcellation methods will be investigated. If successful, the study will: 1) provide a new and effective clinical tool to study plastic cortical changes that occur after SCI, 2) provide a new non-invasive imaging biomarker that is predictive of progress towards recovery in response to therapy, and 3) extend our knowledge about the functional reorganization that takes place during and after therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-65 years) men and women of all ethnic groups
* SCI, traumatic
* Thoracic neurological level, without the involvement of lower motor neurons.
* American Spinal Injury Association (ASIA) classification A-D
* Chronic injury: > 6 months from the injury
* Satisfactory general health
* No FES ergometer (i.e. RT300 or equivalent) use within 4 weeks.
* Ability to comply with procedures and follow-up

Exclusion Criteria:

* Contra-indication to Magnetic Resonance (MR) study (e.g., cardiac pacemaker, claustrophobia, aneurysm clip, etc.)
* History or clinical evidence of moderate or severe brain injury
* Major spine deformity (e.g. scoliosis, kyphosis, subluxation)
* Movement disorder or severe spasticity preventing ability to lay still for extended periods required for imaging.
* Women who are pregnant
* Concurrent lower motor neuron disease such as peripheral neuropathy that would exclude lower extremity electrical excitability
* Unstable long bone fractures of the lower extremities.
* Subjects with history of inability to tolerate electrical stimulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann S Choe, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Kennedy Krieger Institute, International Center for Spinal Cord Injury, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All research material will be kept confidential and any means of subject identification (name and history number) will be removed from all material for analysis or presentation. No identifying information will be made publicly available. In some cases, the study protocol, statistical analysis plan, individual scans, and all Individual Participant Data (IPD) that underlie results in a publication will be included in published papers or meeting papers or posters, but the identity of the subject in question will not be revealed.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Starting immediately after publication
Access Criteria: All IPD that underlie results in a publication will be available to the extent the related publication(s) allows it. However, under no circumstances any IPD that contains subject identification information will be shared.

REFERENCES:
- [Background] Choe AS. Advances in Spinal Functional Magnetic Resonance Imaging in the Healthy and Injured Spinal Cords. Curr Phys Med Rehabil Rep. 2017 Sep;5(3):143-150. doi: 10.1007/s40141-017-0161-x. Epub 2017 Jul 31. PMID 29255645
- [Background] Choe AS, Nebel MB, Barber AD, Cohen JR, Xu Y, Pekar JJ, Caffo B, Lindquist MA. Comparing test-retest reliability of dynamic functional connectivity methods. Neuroimage. 2017 Sep;158:155-175. doi: 10.1016/j.neuroimage.2017.07.005. Epub 2017 Jul 5. PMID 28687517
- [Background] Choe AS, Jones CK, Joel SE, Muschelli J, Belegu V, Caffo BS, Lindquist MA, van Zijl PC, Pekar JJ. Reproducibility and Temporal Structure in Weekly Resting-State fMRI over a Period of 3.5 Years. PLoS One. 2015 Oct 30;10(10):e0140134. doi: 10.1371/journal.pone.0140134. eCollection 2015. PMID 26517540
- [Background] Choe AS, Belegu V, Yoshida S, Joel S, Sadowsky CL, Smith SA, van Zijl PC, Pekar JJ, McDonald JW. Extensive neurological recovery from a complete spinal cord injury: a case report and hypothesis on the role of cortical plasticity. Front Hum Neurosci. 2013 Jun 25;7:290. doi: 10.3389/fnhum.2013.00290. eCollection 2013. PMID 23805087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Started | 9 | 5
Completed | 9 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Functional Electric Stimulation Cycling: The Functional Electrical Stimulation (FES) cycling group will use RT300 ergometer (Restorative Therapies, Inc) with stimulation on.
  Functional Electric Stimulation cycling: The Functional Electrical Stimulation (FES) cycling group will use RT300 ergometer (Restorative Therapies, Inc). Bilateral glutei, quadriceps and hamstrings will be stimulated. The stimulation parameters will be set as follows: waveform biphasic, charged balanced; phase duration of 250 microseconds; pulse rate 33-45 pps. The stimulus intensity will be adjusted for individual patients and muscle group so that a tolerable stimulation is provided that will generate a cycling action. Target cycling speed is 50 RPM. Resistance will be automatically adjusted by the FES bike according to the subject's performance. When fatigue occurs, participants will continue cycling with electrical stimulation and motor support. FES therapy will be administered for one hour per session 3 times a week.
- Total: Total of all reporting groups
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: International Standard of Neurological Classification for Spinal Cord Injury (ISNCSCI) Score
Description: Developed by the American Spinal Injury Association (ASIA), the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) provides an overall assessment of motor and sensory function following spinal cord injury. For this study, a single composite ISNCSCI score is reported, which ranges from 0 (indicating the worst overall function) to 324 (indicating normal overall function). The data table presents this composite score as the sole outcome measure for each Arm/Group.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 9 | 5
score on a scale | 59.5 (11.34) | 60.4 (14.68)

2. Primary Outcome: International Standard of Neurological Classification for Spinal Cord Injury (ISNCSCI) Score
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 7 | 5
score on a scale | 62.2 (15.09) | 61 (15.14)

3. Primary Outcome: International Standard of Neurological Classification for Spinal Cord Injury (ISNCSCI) Score
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 7 | 4
score on a scale | 64.4 (13.49) | 63.5 (14.12)

4. Primary Outcome: Resting State fMRI Functional Connectivity
Description: Resting state functional magnetic resonance imaging (RsfMRI) functional connectivity is defined as the temporal dependency of neuronal activation patterns (represented by the blood oxygenation level dependent (BOLD) signal time courses as measured using rsfMRI) of anatomically separated brain regions. There are number of methodologies one can use to characterize the degree and type of rsfMRI functional connectivity. One example is between-network-connectivity (BNC), which is defined as the degree of correlation between two time courses obtained from a pair of brain regions. Summary statistics of BNC (e.g., mean, variance), as well as the dynamic properties of BNC (e.g., dynamic functional connectivity) can be used to further summarize the characteristics of the functional connectivity in SCI population. Note that the BNC values reported in the Outcome Measure data table represent "Pearson's Correlation Coefficient" and not z-transformed Pearson's Correlation Coefficients.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Unitless (Pearson's correlation coeff)
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 9 | 5
Unitless (Pearson's correlation coeff) | 0.556 (0.152) | 0.587 (0.152)

5. Primary Outcome: Resting State fMRI Functional Connectivity
Description: RsfMRI functional connectivity is defined as the temporal dependency of neuronal activation patterns (represented by the blood oxygenation level dependent (BOLD) signal time courses as measured using rsfMRI) of anatomically separated brain regions. There are number of methodologies one can use to characterize the degree and type of rsfMRI functional connectivity. One example is between-network-connectivity (BNC), which is defined as the degree of correlation between two time courses obtained from a pair of brain regions. Summary statistics of BNC (e.g., mean, variance), as well as the dynamic properties of BNC (e.g., dynamic functional connectivity) can be used to further summarize the characteristics of the functional connectivity in SCI population. Note that the BNC values reported in the Outcome Measure data table represent "Pearson's Correlation Coefficient" and not z-transformed Pearson's Correlation Coefficients.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Unitless (Pearson's correlation coeff)
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 7 | 5
Unitless (Pearson's correlation coeff) | 0.496 (0.119) | 0.493 (0.143)

6. Primary Outcome: Resting State fMRI Functional Connectivity
Description: as for outcome 5
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Unitless (Pearson's correlation coeff)
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 7 | 4
Unitless (Pearson's correlation coeff) | 0.533 (0.120) | 0.496 (0.096)

7. Primary Outcome: Resting-State fMRI Brain Parcels Outcome Measure: Sensorimotor Network (SMN) Recruitment Coefficient
Description: Resting-state functional connectivity can also identify functionally homogeneous brain regions, or "parcels." By examining each parcel's properties, such as the center of mass and recruitment coefficient value, we can gain insights into the brain's functional reorganization. Given its importance in the SCI population, we focused on the sensorimotor network (SMN) parcel.
  RsfMRI data were collected and preprocessed. The brain data was then parcellated into 200 parcels. Next, a multi-layer community detection algorithm was applied to identify cohesive subnetworks over time, and the SMN Recruitment Coefficient was calculated - which is a dimensionless metric that quantifies how strongly the SMN parcels cohere, or preferentially connect, with one another compared to parcels in other networks. Higher values suggest a more internally cohesive SMN, indicating stronger functional segregation and potentially more intact sensorimotor function.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Unitless coefficient (dimensionless)
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 9 | 5
Unitless coefficient (dimensionless) | 0.491 (0.0880) | 0.4670 (0.0914)

8. Primary Outcome: Resting-State fMRI Brain Parcels Outcome Measure: Sensorimotor Network (SMN) Recruitment Coefficient
Description: as for outcome 7
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Unitless coefficient (dimensionless)
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 7 | 5
Unitless coefficient (dimensionless) | 0.813 (0.119) | 0.484 (0.0737)

9. Primary Outcome: Resting-State fMRI Brain Parcels Outcome Measure: Sensorimotor Network (SMN) Recruitment Coefficient
Description: as for outcome 7
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Unitless coefficient (dimensionless)
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
Number analyzed (Participants) | 7 | 4
Unitless coefficient (dimensionless) | 0.713 (0.146) | 0.581 (0.102)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Functional Electric Stimulation Cycling | Passive Cycling
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03854214/Prot_SAP_000.pdf